CLINICAL TRIAL: NCT03617224
Title: Phase I Trial of Pembrolizumab and Total Skin Electron Beam Radiotherapy in Mycosis Fungoides and Sézary Syndrome
Brief Title: Pembrolizumab and Total Skin Electron Beam Radiotherapy in Mycosis Fungoides and Sézary Syndrome
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to enroll patients that met enrollment criteria.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 032018-018
Record Dates: First submitted 2018-07-27; First posted 2018-08-06 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Cutaneous T-Cell Lymphomas
Keywords: Mycosis Fungoides (MF), Sezary Syndrome (SS), Pembrolizumab, Total Skin Electron Beam Therapy (TSEBT)
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TSEBT and pembrolizumab (Experimental): Dose regimens are sequential therapy of TSEBT with Pembrolizumab.
  Interventions: Drug: TSEBT and pembrolizumab
- Radiation: TSEBT (Experimental): The regimen includes a rule-based "3+3" design for escalating regimen intensity of combined TSEBT and pembrolizumab.
  Interventions: Radiation: TSEBT

INTERVENTIONS:
Radiation: TSEBT — The regimen includes a rule-based "3+3" design for escalating regimen intensity of combined TSEBT and pembrolizumab.
  Arms: Radiation: TSEBT
Drug: TSEBT and pembrolizumab — Dose regimens are sequential therapy of TSEBT with Pembrolizumab.
  Arms: TSEBT and pembrolizumab

SUMMARY:
Hypothesis: Addition of low dose TSEBT to debulk MF/SS either before or during checkpoint blockade with anti-PD-1 pembrolizumab monoclonal antibody therapy will be safe and well tolerated.

Primary Objective:

• To determine the maximum tolerated dose (MTD) for the combination of total skin electron beam therapy (TSEBT) and pembrolizumab regimen.

Secondary Objectives:

* To determine the preliminary efficacy of the combination of TSEBT with pembrolizumab.
* To determine the impact on patient-reported health-related quality of life outcomes.

DETAILED DESCRIPTION:
This is a single center phase I clinical trial assessing the safety of combination therapy of TSEBT and pembrolizumab for treatment of Stage IB-IV relapsed/refractory MF and SS.

Primary Endpoint:

• Primary endpoint will be maximum tolerated dose (MTD).

Secondary Endpoints:

* Efficacy of the combination of TSEBT with pembrolizumab therapy is measured.
* CTCAE v4.0 toxicity beyond the 30 day period following the second therapy in the combination protocol treatment and up to 30 days following last dose of pembrolizumab.
* Skindex-29 patient-reported HRQOL survey.

Sample Size and Accrual: 18 patients will be enrolled.

Statistical Analysis: Time to event will be estimated using the Kaplan-Meier approach along with the 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed Mycosis Fungoides or Sézary Syndrome
* Stage IB-IV by ISCL/EORTC 2007 Revision Staging (See Appendix Section 13.3). Maximal stage since diagnosis will determine eligibility.
* Failed or intolerant to at least one prior line of systemic therapy
* Life expectancy > 6 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2 and able to stand for TSEBT
* Baseline measurable disease by the mSWAT criteria
* Acceptable baseline laboratories:

  * Leukocytes ≥ 2,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcl
  * Hemoglobin ≥ 9g/dL
  * Total bilirubin ≤ 1.5 X institutional upper limit of normal
  * AST(SGOT)/ALT(SPGT) ≤ 2.5 X institutional upper limit of normal
  * INR/PT ≤ 1.5 X institutional upper limit of normal (*unless on anticoagulation therapy and therapeutic)
  * Serum creatinine ≤ 1.5 X institutional upper limit normal OR ≥ 60 mL/min calculated creatinine clearance ≥60 mL/min for subject
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent.
* Patient must provide tissue biopsy (punch) of skin at baseline (pre-study treatment), following 3 cycles of pembrolizumab, 1 month following end of TSEBT, at clinical event of progression, at end of treatment (unless at same time as progression triggered biopsy). Optional biopsy can be taken every 3 cycles of pembrolizumab and at time of initial response to pembrolizumab.
* Must be a candidate for TSEBT

Exclusion Criteria:

* Subjects who have had prior TSEBT (prior focal radiotherapy is allowed).
* Subjects who have had systemic cytotoxic anticancer agents or radiotherapy within 2 weeks prior to entering the study or those who have not in the opinion of the treating physician recovered from adverse events due to agents administered more than 2 weeks earlier.
* Subjects who have received the following prior therapies:
* Alemtuzumab within the past 8 weeks
* Retinoids, interferons, Vorinostat, Romidepsin, oral corticosteroids (except physiologic replacement dose or topicals) within the past 2 weeks
* Phototherapy within the past 4 weeks
* Topical therapies including retinoids, nitrogen mustards and Imiquimod within the past week
* Patients may not have received systemic steroid therapy or other form of immunosuppressive therapy within 7 days prior to the first dose of pembrolizumab
* Subjects may not be receiving any other investigational agents during the study or for within 4 weeks of registration.
* Subjects with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Subjects with known history of immunodeficiency or severe autoimmune disease requiring systemic immunosuppressive agents or severe connective tissue diseases (i.e. systemic scleroderma) or DNA damage repair deficiency syndromes that are known to pre-dispose to excess DNA damage hypersensitivity from ionizing radiation will be excluded from the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active hepatitis B or C, history of pneumonitis requiring steroids, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects must not have received a recent live vaccine within 30 days of treatment.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Patients with history of hypersensitivity to monoclonal antibodies.
* History of prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-3475 (pembrolizumab)
* Patients may not have an additional known malignancy requiring active treatment or which his progressing, excluding non-melanoma skin cancer or in situ cervical cancer which has undergone potentially curative therapy.
* Known human T-lymphotropic virus type 1 (HTLV) infection
* History of non-infectious pneumonitis requiring steroids

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2022-07-24 (Estimated); Study Completion 2024-07-24 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 1 Year
  The highest dose in the regimen is assessed if dose limiting toxicities do not halt escalation.

SECONDARY OUTCOMES:
Response to therapy | 4 Years
  The response to therapy is measured from overall response criteria from initiation of any therapy.
Progression-free survival | 4 Years
  Progression-free survival is measured without the development of new metastasis.
Health-related quality of life (HRQOL) | 4 Years
  HRQOL's are measured using the Skindex-29. The higher the number better the quality of life.
Dose Limiting Toxicities (DLT) | 4 Years
  Severity or Toxicity will be assessed according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0. Dose adjustments should be made according to the system showing the greatest degree of toxicity. The consequences of toxicity should all be graded 1-5 according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 occurring prior to 270 days from the start of protocol treatment. CTCAE V4.0 along with grades 1-5 is provided in the link for reference (https://evs.nci.nih.gov/ftp1/CTCAE/CTCAE_4.03/CTCAE_4.03_2010-06 14_QuickReference_8.5x11.pdf).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No